CLINICAL TRIAL: NCT00149175
Title: Clinical and Genetic Study of Neurodegenerative Disorders With Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: RBM02-59; DGS2004/0525 (Registry Identifier: Reference DGS)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease; Dementia; Neurodegenerative Disorders
Keywords: Alzheimer's disease; Dementia; Phenotype-genotype correlations; Candidate genes; Related disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Neurodegenerative disorders with cognitive impairment
  Interventions: Other: Blood sampling, skin biopsy
- Control
  Interventions: Other: Blood sampling, skin biopsy
- At risk reactive
  Interventions: Other: Blood sampling, skin biopsy

INTERVENTIONS:
Other: Blood sampling, skin biopsy — Blood sampling, skin biopsy in the field of the medical follow-up

SUMMARY:
Patients with different types of dementia will be recruited and evaluated in national hospital departments for their usual neurological follow-ups. A blood sample will be proposed in the field of this research project, and the biological material will be stored at the DNA and Cell Bank of Institut de Fédératif Recherche (IFR) of Neurosciences (Pitié-Salpêtrière Hospital, Paris). The clinical research network is already set up for Alzheimer's disease and frontotemporal dementias, which permits an evaluation according to a clinical standardized protocol.

Among these disorders, a monogenic sub-group has been identified. In Alzheimer's disease, it is associated with the APP, PSEN1 and PSEN2 genes, which account only for 75% of the familial forms with early onset. In frontotemporal dementias, the tau gene mutations account only for 10% of the cases with an autosomal dominant inheritance. The identification of familial forms with a genetic inquiry in the relatives is essential for a greater knowledge of the molecular bases of forms not caused by the known genes, using linkage approaches and candidate gene analysis. The familial forms are also useful for identifying the modifier genes.

In the multifactorial forms, the aim is to assemble a wide cohort of patients and controls matched for localizing and identifying susceptibility genetic factors. The strategies will use a candidate gene approach, and in the near future, studies of single nucleotide polymorphisms (SNPs) spread out in the whole genome. Meanwhile, similar approaches, particularly with candidate genes, could be used for identifying predictive factors of tolerance and response to the treatment.

Finally, correlations will be performed with seric markers according to each kind of dementia.

Specialized clinical teams in diagnosis and follow-up in dementias are assembled for this project, and in the study of neurological disorders of genetic origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with a neurodegenerative disorder with cognitive impairment controls (without signs of the disease), matched with sex and age with the patients
* Relatives for the familial cases

Exclusion Criteria:

* Pregnant women
* Minors
* Persons refusing to sign the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients presenting with a neurodegenerative disorder
  * At risk patients
Sampling Method: Non-Probability Sample
Enrollment: 2256 (Actual)
Dates: Start 2002-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Brice, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, University Paris 6
Locations (12):
- France (12):
  - CHU de la Côte de Nacre, Caen
  - Hôpital Sainte-Marguerite, Marseille
  - Hôpital Guillaume et René Laennec, Nantes
  - Hôpital de l'Archet, Nice
  - Pitié-Salpêtrière Hospital - Centre du Langage et de Neuropsychologie, Paris
  - Pitié-Salpêtrière Hospital - Fédération de Neurologie, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Centre Hospitalier, Saint-Brieuc
  - Hôpital Bellevue, Saint-Etienne
  - Hôpital Civil, Strasbourg

REFERENCES:
- [Background] Le Ber I, Guedj E, Gabelle A, Verpillat P, Volteau M, Thomas-Anterion C, Decousus M, Hannequin D, Vera P, Lacomblez L, Camuzat A, Didic M, Puel M, Lotterie JA, Golfier V, Bernard AM, Vercelletto M, Magne C, Sellal F, Namer I, Michel BF, Pasquier J, Salachas F, Bochet J; French research network on FTD/FTD-MND; Brice A, Habert MO, Dubois B. Demographic, neurological and behavioural characteristics and brain perfusion SPECT in frontal variant of frontotemporal dementia. Brain. 2006 Nov;129(Pt 11):3051-65. doi: 10.1093/brain/awl288. PMID 17071924
- [Background] van der Zee J, Le Ber I, Maurer-Stroh S, Engelborghs S, Gijselinck I, Camuzat A, Brouwers N, Vandenberghe R, Sleegers K, Hannequin D, Dermaut B, Schymkowitz J, Campion D, Santens P, Martin JJ, Lacomblez L, De Pooter T, Peeters K, Mattheijssens M, Vercelletto M, Van den Broeck M, Cruts M, De Deyn PP, Rousseau F, Brice A, Van Broeckhoven C. Mutations other than null mutations producing a pathogenic loss of progranulin in frontotemporal dementia. Hum Mutat. 2007 Apr;28(4):416. doi: 10.1002/humu.9484. PMID 17345602
- [Background] Baba Y, Baker MC, Le Ber I, Brice A, Maeck L, Kohlhase J, Yasuda M, Stoppe G, Bugiani O, Sperfeld AD, Tsuboi Y, Uitti RJ, Farrer MJ, Ghetti B, Hutton ML, Wszolek ZK. Clinical and genetic features of families with frontotemporal dementia and parkinsonism linked to chromosome 17 with a P301S tau mutation. J Neural Transm (Vienna). 2007 Jul;114(7):947-50. doi: 10.1007/s00702-007-0632-9. Epub 2007 Feb 23. PMID 17318302
- [Background] Le Ber I, van der Zee J, Hannequin D, Gijselinck I, Campion D, Puel M, Laquerriere A, De Pooter T, Camuzat A, Van den Broeck M, Dubois B, Sellal F, Lacomblez L, Vercelletto M, Thomas-Anterion C, Michel BF, Golfier V, Didic M, Salachas F, Duyckaerts C, Cruts M, Verpillat P, Van Broeckhoven C, Brice A; French Research Network on FTD/FTD-MND. Progranulin null mutations in both sporadic and familial frontotemporal dementia. Hum Mutat. 2007 Sep;28(9):846-55. doi: 10.1002/humu.20520. PMID 17436289
- [Background] Guedj E, Le Ber I, Lacomblez L, Dubois B, Verpillat P, Didic M, Salachas F, Vera P, Hannequin D, Lotterie JA, Puel M, Decousus M, Thomas-Anterion C, Magne C, Vercelletto M, Bernard AM, Golfier V, Pasquier J, Michel BF, Namer I, Sellal F, Bochet J, Volteau M, Brice A, Meininger V; French Research Network on FTD/FTD-MND; Habert MO. Brain spect perfusion of frontotemporal dementia associated with motor neuron disease. Neurology. 2007 Jul 31;69(5):488-90. doi: 10.1212/01.wnl.0000266638.53185.e7. No abstract available. PMID 17664410
- See also: Related Info — http://www.inserm.fr